CLINICAL TRIAL: NCT04472598
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study Of Navitoclax In Combination With Ruxolitinib Versus Ruxolitinib In Subjects With Myelofibrosis (TRANSFORM-1)
Brief Title: Study of Oral Navitoclax Tablet In Combination With Oral Ruxolitinib Tablet When Compared With Oral Ruxolitinib Tablet To Assess Change In Spleen Volume In Adult Participants With Myelofibrosis
Acronym: TRANSFORM-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-191; 2020-000097-15 (EudraCT Number)
Expanded Access: NCT03592576 (No longer available)
Record Dates: First submitted 2020-07-14; First posted 2020-07-15 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Myelofibrosis (MF)
Keywords: Myelofibrosis; Navitoclax; Ruxolitinib; Cancer; ABT-263; TRANSFORM-1
MeSH Terms: conditions — Primary Myelofibrosis; Neoplasms | interventions — navitoclax; ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Navitoclax + Ruxolitinib (Experimental): Participants will receive Navitoclax in combination with Ruxolitinib
  Interventions: Drug: Navitoclax; Drug: Ruxolitinib
- Placebo for Navitoclax + Ruxolitinib (Active Comparator): Participants will receive placebo for Navitoclax and Ruxolitinib
  Interventions: Drug: Ruxolitinib; Drug: Placebo for Navitoclax

INTERVENTIONS:
Drug: Navitoclax — Tablet; Oral
  Other Names: ABT-263
  Arms: Navitoclax + Ruxolitinib
Drug: Ruxolitinib — Tablet; Oral
Drug: Placebo for Navitoclax — Tablet; Oral
  Arms: Placebo for Navitoclax + Ruxolitinib

SUMMARY:
Myelofibrosis is a type of bone marrow cancer that usually develops slowly and disrupts body's normal production of blood cells. It causes bone marrow scarring, leading to severe anemia that can cause weakness and fatigue. It can also cause a low number of blood-clotting cells called platelets, which increases risk of bleeding. Myelofibrosis often causes an enlarged spleen. The purpose of this study is to see if a combination of navitoclax and ruxolitinib is more effective and safe in assessment of change in spleen volume when compared to ruxolitinib in participants with myelofibrosis.

Navitoclax is an investigational drug for the treatment of myelofibrosis. Participants in this study are divided into two groups, called treatment arms. Each group receives a different treatment. Adult participants with a diagnosis of myelofibrosis will be enrolled. Around 230 participants will be enrolled in approximately 190 sites worldwide.

Participants will receive oral navitoclax tablet with oral ruxolitinib tablet or oral ruxolitinib tablet with oral placebo (no active drug) tablet and treatment may continue untill the participant cannot tolerate the study drug, or benefit is not achieved, or other reasons which qualify for discontinuation of the study drug.

There may be a higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, magnetic resonance imaging (MRI) or computed tomography (CT) scan, bone marrow tests, checking for side effects, and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of Primary MyeloFibrosis (MF) as defined by World Health Organization (WHO) classification or Secondary MF (post polycythemia vera [PPV] - MF or Post Essential Thrombocytopenia [PET] - MF) .
* Must be able to complete the MF Symptom Assessment Form (MFSAF) v4.0 on at least 4 out of 7 days immediately preceding the date of randomization.

  -- Must have at least 2 symptoms with a score >=3 or a total score of >=12, as measured by the MFSAF v4.0.
* Classified as intermediate-2, or high-Risk MF as defined by the Dynamic International Prognostic Scoring System Plus (DIPSS+).
* Has splenomegaly defined as spleen palpation measurement >= 5 centimeters (cm) below costal margin or spleen volume greater than or equal to 450 cubic cm as assessed centrally by magnetic resonance imaging (MRI) or computed tomography (CT) scan.
* Ineligible for stem cell transplantation at time of study entry due to age, comorbidities, or unfit for unrelated or unmatched donor transplant and other criteria per National Comprehensive Cancer Network guidelines.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.

Exclusion Criteria:

* Prior treatment with a Janus Kinase-2 (JAK-2) inhibitor.
* Prior treatment with a B-cell lymphoma 2 homology 3 (BH3)-mimetic compound or bromodomain and extra-terminal motif (BET) inhibitor or stem cell transplant.
* Receiving medication that interferes with coagulation or platelet function within 3 days prior to the first dose of study drug or during the study treatment period except for low dose aspirin (up to 100 milligram daily) and low molecular weight heparin (LMWH).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who achieve Spleen Volume Reduction of at least 35% at Week 24 (SVR35W24) | At Week 24
  Reduction in spleen volume is measured by magnetic resonance imaging (MRI) or computed tomography (CT), per International Working Group (IWG) criteria.

SECONDARY OUTCOMES:
Change in Total Symptom Score (TSS) | Baseline (Week 0) Up to Week 24
  Reduction in TSS is measured by Myelofibrosis Symptom Assessment Form (MFSAF) v4.0.
Percentage of Participants who achieve Spleen Volume Reduction of at least 35% (SVR35) | Baseline (Week 0) Up to Week 96
  Reduction in spleen volume is measured by MRI or CT, per IWG criteria.
Duration of 35% Spleen Volume Reduction (SVR35) | Baseline (Week 0) Up to Week 96
  Duration of SVR35 is defined as the time between the date of first response of spleen volume reduction of 35% achievement to the date of the first assessment where the spleen volume is less than 35% reduction from baseline and is at least 25% increase from the nadir (the lowest spleen volume).
Change In Fatigue | Baseline (Week 0) Up to Week 24
  Change in fatigue will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue SF 7a.
Change in Physical Functioning | Baseline (Week 0) Up to Week 24
  Change in physical functioning is measured by the physical functioning domain of the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 or death.
Percentage of Participants who achieve Anemia Response | Baseline (Week 0) Up to Week 96
  The rate of anemia response will be assessed according to current International Working Group-Myeloproliferative Neoplasms Research and European LeukemiaNet (IWG-MRT/ELN) criteria.
Overall Survival (OS) | Up To approximately 8 Years
  OS is defined as the time from the date of randomization to the date of death from any cause.
Leukemia-Free Survival | Up To approximately 8 Years
  Leukemia-free survival is defined as the number of days from the date of randomization to the onset date of documented leukemia, disease progression due to leukemia, or death due to leukemia, whichever occurs first.
Percentage of Participants who Achieve Reduction in Grade of Bone Marrow Fibrosis | Baseline (Week 0) Up to Week 96
  Change in grade of bone marrow fibrosis will be measured per the European consensus grading system through bone marrow biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (194):
- United States (35):
  - Highlands Oncology Group, PA /ID# 221824, Springdale, Arkansas
  - Providence - St. Jude Medical Center /ID# 241646, Fullerton, California
  - Moores Cancer Center at UC San Diego /ID# 218012, La Jolla, California
  - Rocky Mountain Cancer Centers - Littleton /ID# 222562, Littleton, Colorado
  - Lynn Cancer Institute, Boca /ID# 230687, Boca Raton, Florida
  - Florida Cancer Specialist - South /ID# 221726, Fort Myers, Florida
  - Florida Cancer Specialists - North /ID# 221727, St. Petersburg, Florida
  - Florida Cancer Specialists - East /ID# 221728, West Palm Beach, Florida
  - Emory University /ID# 221562, Atlanta, Georgia
  - Augusta University Georgia Cancer Center /ID# 221551, Augusta, Georgia
  - Columbus Regional Research Institute /ID# 227272, Columbus, Georgia
  - Duplicate_Rush University Medical Center /ID# 221581, Chicago, Illinois
  - Mid Illinois Hematology & Oncology Associates, Ltd /ID# 224204, Normal, Illinois
  - Indiana Blood & Marrow Transpl /ID# 221586, Indianapolis, Indiana
  - University of Kansas Cancer Center /ID# 218144, Fairway, Kansas
  - Massachusetts General Hospital /ID# 221559, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center /ID# 224261, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 218010, Boston, Massachusetts
  - University of Michigan /ID# 221658, Ann Arbor, Michigan
  - Minnesota Oncology Hematology /ID# 227357, Edina, Minnesota
  - MidAmerica Division, Inc. /ID# 221743, Kansas City, Missouri
  - Hackensack Univ Med Ctr /ID# 221654, Hackensack, New Jersey
  - Northwell Health - Monter Cancer Center /ID# 222996, Lake Success, New York
  - Weill Cornell Medical College /ID# 220933, New York, New York
  - Gabrail Cancer Center Research /ID# 230488, Canton, Ohio
  - Oncology Hematology Care, Inc. /ID# 222556, Cincinnati, Ohio
  - The Ohio State University /ID# 221584, Columbus, Ohio
  - UPMC Hillman Cancer Ctr /ID# 218134, Pittsburgh, Pennsylvania
  - Thompson Cancer Survival Ctr /ID# 231689, Knoxville, Tennessee
  - University of Texas MD Anderson Cancer Center /ID# 217994, Houston, Texas
  - Texas Oncology - Northeast Texas /ID# 241813, Tyler, Texas
  - Utah Cancer Specialists Salt Lake Clinic /ID# 221961, Salt Lake City, Utah
  - University of Utah /ID# 221009, Salt Lake City, Utah
  - Virginia Cancer Specialists - Fairfax /ID# 242682, Fairfax, Virginia
  - VA Puget Sound Health Care System /ID# 231691, Seattle, Washington
- Australia (8):
  - The Kinghorn Cancer Centre /ID# 221503, Darlinghurst, New South Wales
  - Border Medical Oncology Research Unit Albury Wodonga Regiona /ID# 231311, East Albury, New South Wales
  - Gosford Hospital /ID# 221499, Gosford, New South Wales
  - Liverpool Hospital /ID# 221803, Liverpool, New South Wales
  - Townsville University Hospital /ID# 229794, Douglas, Queensland
  - Peter MacCallum Cancer Ctr /ID# 229795, Melbourne, Victoria
  - The Alfred Hospital /ID# 221501, Melbourne, Victoria
  - Royal Perth Hospital /ID# 223203, Perth, Western Australia
- Austria (5):
  - Duplicate_Medizinische Universitaet Graz /ID# 220910, Graz, Styria
  - Ordensklinikum Linz GmbH Elisabethinen /ID# 220813, Linz, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH /ID# 220901, Wels, Upper Austria
  - Medizinische Universitaet Wien /ID# 220906, Vienna, Vienna
  - Hanusch Krankenhaus /ID# 220909, Vienna
- Belgium (8):
  - ZAS Cadix /ID# 221465, Antwerp, Antwerpen
  - CHU de Liège /ID# 218874, Liège, Liege
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant /ID# 221127, Yvoir, Namur
  - UZ Gent /ID# 221125, Ghent, Oost-Vlaanderen
  - Vitaz /Id# 229861, Sint-Niklaas, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 218806, Leuven, Vlaams-Brabant
  - AZ-Delta /ID# 221466, Roeselare, West-Vlaanderen
  - AZ Sint-Jan Brugge /ID# 218805, Bruges
- Bulgaria (5):
  - UMHAT Alexandrovska EAD /ID# 231056, Sofiya, Sofia
  - UMHAT Dr Georgi Stranski EAD /ID# 231161, Pleven
  - UMHAT Sveti Georgi /ID# 231053, Plovdiv
  - Acibadem City Clinic Tokuda University Hospital EAD /ID# 231036, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 231028, Sofia
- Canada (5):
  - Royal Victoria Hospital /ID# 222636, Barrie, Ontario
  - Juravinski Cancer Centre /ID# 221752, Hamilton, Ontario
  - Lakeridge Health - Oshawa /ID# 222080, Oshawa, Ontario
  - Niagara Health System /ID# 230994, St. Catharines, Ontario
  - CHUQ- Hôpital de l'Enfant-Jesus /ID# 221754, Québec, Quebec
- Croatia (4):
  - Clinical Hospital Dubrava /ID# 230795, Zagreb, City of Zagreb
  - Klinicka bolnica Merkur /ID# 231155, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 230793, Zagreb, City of Zagreb
  - Duplicate_Klinicki bolnicki centar Split /ID# 230796, Split, Split-Dalmatia County
- France (11):
  - CHU NIMES - Hopital Caremeau /ID# 219114, Nîmes, Gard
  - Centre Hospitalier Universitaire de Bordeaux /ID# 222518, Pessac, Gironde
  - CH Roubaix - Hopital Victor Provo /ID# 219116, Roubaix, Hauts-de-France
  - CHU de Nantes, Hotel Dieu -HME /ID# 219113, Nantes, Pays de la Loire Region
  - HCL - Hopital Lyon Sud /ID# 222913, Pierre-Bénite, Rhone
  - Centre Hospitalier Métropole Savoie - Site Hôpital de Chambéry /ID# 224506, Chambéry, Savoie
  - Chu Angers /Id# 219115, Angers
  - Hôpital Saint-Louis /ID# 221288, Paris
  - AP-HP - Hopital Necker /ID# 231318, Paris
  - ICANS - Institut de Cancérologie Strasbourg Europe /ID# 229978, Strasbourg
  - Hopital Avicenne - APHP /ID# 221286, Bobigny, Île-de-France Region
- Germany (7):
  - Universitatsklinikum Mannheim /ID# 221523, Mannheim, Baden-Wurttemberg
  - Haemato-Onkologie /ID# 221061, Munich, Bavaria
  - Universitaetsklinikum Aachen /ID# 221519, Aachen, North Rhine-Westphalia
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf /ID# 221347, Dresden, Saxony
  - Universitaetsklinikum Essen /ID# 221522, Essen
  - OncoResearch Lerchenfeld GmbH /ID# 230867, Hamburg
  - Klinikum rechts der Isar /ID# 221520, Munich
- Greece (3):
  - General Hospital of Athens Laiko /ID# 230785, Athens, Attica
  - Duplicate_University General Hospital Attikon /ID# 230784, Athens, Attica
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 230786, Athens
- Israel (6):
  - Meir Medical Center /ID# 221374, Kfar Saba, Central District
  - Yitzhak Shamir Medical Center /ID# 222957, Ẕerifin, Central District
  - Rambam Health Care Campus /ID# 219120, Haifa, H_efa
  - Hadassah Medical Center-Hebrew University /ID# 219110, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 219137, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 219134, Tel Aviv, Tel Aviv
- Italy (7):
  - IRCCS AOU di Bologna - Policlinico Sant'Orsola-Malpighi /ID# 220867, Bologna, Emilia-Romagna
  - Azienda Ospedaliero Universitaria Careggi /ID# 219086, Florence, Firenze
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 219083, Rome, Roma
  - ASST Papa Giovanni XXIII /ID# 221907, Bergamo
  - ASST degli Spedali Civili di Brescia /ID# 241273, Brescia
  - AOU Policlinico G. Rodolico - San Marco /ID# 219085, Catania
  - Duplicate_ASST Sette Laghi /ID# 219084, Varese
- Japan (28):
  - Japanese Red Cross Aichi Medical Center Nagoya Daiichi Hospital /ID# 239100, Nagoya, Aichi-ken
  - Fujita Health University Hospital /ID# 221537, Toyoake, Aichi-ken
  - Duplicate_Chiba University Hospital /ID# 239345, Chiba, Chiba
  - National Cancer Center Hospital East /ID# 226093, Kashiwa-shi, Chiba
  - Ehime University Hospital /ID# 221443, Toon-shi, Ehime
  - Kyushu University Hospital /ID# 221783, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital /ID# 222752, Fukushima, Fukushima
  - Ogaki Municipal Hospital /ID# 240173, Ogaki-shi, Gifu
  - Gunmaken Saiseikai Maebashi Hospital /ID# 242806, Maebashi, Gunma
  - Gunma University Hospital /ID# 221480, Maebashi, Gunma
  - Duplicate_Hokkaido University Hospital /ID# 242667, Sapporo, Hokkaido
  - Kobe University Hospital /ID# 246236, Kobe, Hyōgo
  - Hitachi General Hospital /ID# 240048, Hitachi-shi, Ibaraki
  - Kanazawa University Hospital /ID# 238424, Kanazawa, Ishikawa-ken
  - Medical Corporation Seijinkai Ikeda Hospital /ID# 242172, Kanoya-shi, Kagoshima-ken
  - Kyoto University Hospital /ID# 238423, Kyoto, Kyoto
  - Mie University Hospital /ID# 221664, Tsu, Mie-ken
  - University of Miyazaki Hospital /ID# 221483, Miyazaki, Miyazaki
  - Duplicate_Kawasaki Medical School Hospital /ID# 221481, Kurashiki-shi, Okayama-ken
  - Kurashiki Central Hospital /ID# 221692, Kurashiki-shi, Okayama-ken
  - Kansai Medical University Hospital /ID# 221482, Hirakata-shi, Osaka
  - Kindai University Hospital /ID# 221479, Osakasayama-shi, Osaka
  - Osaka University Hospital /ID# 221478, Suita-shi, Osaka
  - Dokkyo Medical University Saitama Medical Center /ID# 222333, Koshigaya, Saitama
  - Juntendo University Shizuoka Hospital /ID# 221782, Izunokuni-shi, Shizuoka
  - Juntendo University Hospital /ID# 221405, Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital /ID# 221674, Bunkyo-ku, Tokyo
  - University of Yamanashi Hospital /ID# 221701, Chuo-shi, Yamanashi
- Netherlands (4):
  - Radboud Universitair Medisch Centrum /ID# 218948, Nijmegen, Gelderland
  - Albert Schweitzer Ziekenhuis /ID# 224015, Dordrecht, South Holland
  - Universitair Medisch Centrum Groningen /ID# 218947, Groningen
  - Universitair Medisch Centrum Utrecht /ID# 218949, Utrecht
- Aotearoa Clinical Trials /ID# 230770, Papatoetoe, Auckland, New Zealand
- Russia (7):
  - Moscow State budget healthcare /ID# 221025, Moscow, Moscow
  - Republican hospital named after V.A. Baranov /ID# 221412, Petrozavodsk, Murmansk Oblast
  - Clinic UZI 4D /ID# 221024, Pyatigorsk, Stavropol Kray
  - Russian Research Institute of Hematology and Transfusiology of the FMBA /ID# 221029, Saint Petersburg
  - Leningrad Regional Clinical Hospital /ID# 221028, Saint Petersburg
  - Almazov National Medical Research Centre /ID# 221033, Saint Petersburg
  - Tula Regional Clinical Hospital /ID# 221027, Tula
- Serbia (4):
  - University Clinical Center Serbia /ID# 230854, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 230946, Belgrade, Beograd
  - University Clinical Center Kragujevac /ID# 230855, Kragujevac, Pomoravski Okrug
  - Duplicate_Clinical Center Vojvodina /ID# 230853, Novi Sad, Vojvodina
- South Africa (3):
  - Wits Clinical Research /ID# 232072, Johannesburg, Gauteng
  - Duplicate_Wits Clinical Research Site /ID# 232071, Johannesburg, Gauteng
  - Alberts Cellular Therapy /ID# 232073, Pretoria, Gauteng
- South Korea (9):
  - Duplicate_Inje University Busan Paik Hospital /ID# 231667, Busan, Busan Gwang Yeogsi
  - Pusan National University Hospital /ID# 222087, Busan, Busan Gwang Yeogsi
  - Duplicate_Kyungpook National University Hospital /ID# 231666, Daegu, Daegu Gwang Yeogsi
  - Gachon University Gil Medical Center /ID# 222089, Incheon, Gyeonggido
  - Duplicate_Seoul National University Bundang Hospital /ID# 219053, Seongnam, Gyeonggido
  - Seoul National University Hospital /ID# 219055, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 219054, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 221068, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 219056, Seoul, Seoul Teugbyeolsi
- Spain (11):
  - Duplicate_Hospital Clínico Universitario de Santiago-CHUS /ID# 222264, Santiago de Compostela, A Coruna
  - Hospital Universitario Germans Trias i Pujol /ID# 229936, Badalona, Barcelona
  - Hospital Universitario Dr. Negrin /ID# 220897, Las Palmas de Gran Canaria, Las Palmas
  - Clinica Universidad de Navarra - Pamplona /ID# 230720, Pamplona, Navarre
  - Hospital Parc de Salut del Mar /ID# 220913, Barcelona
  - Hospital Universitario Vall d'Hebron /ID# 229690, Barcelona
  - CLINICA UNIVERSIDAD DE NAVARRA-Madrid /ID# 230721, Madrid
  - Hospital Universitario Ramon y Cajal /ID# 220877, Madrid
  - Hospital Universitario 12 de Octubre /ID# 229691, Madrid
  - Hospital Universitario Virgen de la Victoria /ID# 220878, Málaga
  - Hospital Clinico Universitario de Valencia /ID# 220875, Valencia
- Sweden (3):
  - Duplicate_Skane University Hospital Lund /ID# 220835, Lund, Skåne County
  - Duplicate_Sahlgrenska University Hospital /ID# 218776, Gothenburg, Västra Götaland County
  - Orebro Universitetssjukhuset /ID# 220829, Örebro, Örebro County
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 218984, Kaohsiung City, Kaohsiung
  - Chi Mei Hospital - Liouying /ID# 221145, Tainan, Tainan
  - National Taiwan University Hospital /ID# 218976, Taipei City, Taipei
  - China Medical University Hospital /ID# 218978, Taichung
  - Taipei Veterans General Hosp /ID# 221146, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 218983, Taoyuan
- Turkey (Türkiye) (5):
  - Hacettepe University Medical Faculty /ID# 230759, Ankara
  - Trakya University Medical Facu /ID# 230754, Edirne, Istanbul
  - Bagcilar Medipol Mega Universite Hastanesi /ID# 230757, Istanbul
  - Ege University Medical Faculty /ID# 230753, Izmir
  - Inonu University Medical Faculty /ID# 230758, Malatya
- Ukraine (4):
  - Communal non-profit enterprise Regional Center of Oncology /ID# 230832, Kharkiv, Kharkivs’ka Oblast’
  - Medical Center OK Clinic LLC, International Institute of Clinical Research /ID# 230834, Kyiv
  - Feofaniya Clinical Hospital of State Management of Affairs /ID# 232370, Kyiv
  - SI Institute of Blood Pathology and Transfusion Medicine of NAMS of Ukraine /ID# 230833, Lviv
- United Kingdom (5):
  - Guys and St Thomas NHS Foundation Trust /ID# 219185, London, Greater London
  - United Lincolnshire Hospitals NHS Trust /ID# 231471, Lincoln, Lincolnshire
  - Oxford University Hospitals NHS Foundation Trust /ID# 219192, Oxford, Oxfordshire
  - University Hospitals Birmingham NHS Foundation Trust /ID# 221333, Birmingham
  - The Christie Hospital /ID# 219191, Manchester

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M16-191